CLINICAL TRIAL: NCT02703870
Title: Combined tDCS and Vision Restoration Training in Post-acute Stroke: an Exploratory Efficacy and Safety Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Magdeburg (Other)
Collaborators: Neurologisches Therapiezentrum Gmundnerberg (Other)
Responsible Party: Principal Investigator, Bernhard A. Sabel, Prof. Dr., University of Magdeburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CES_NTG_1
Record Dates: First submitted 2015-09-18; First posted 2016-03-09 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Hemianopia; Stroke
MeSH Terms: conditions — Hemianopsia; Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Verum tDCS (Active Comparator): Verum group receiving complete treatment of tDCS
  Interventions: Device: verum tDCS; Behavioral: VRT
- sham tDCS (Sham Comparator): Sham group receiving sham tDCS
  Interventions: Device: sham tDCS; Behavioral: VRT
- real VRT (Active Comparator): Real Vision Restoration Training
  Interventions: Device: verum tDCS; Device: sham tDCS

INTERVENTIONS:
Device: verum tDCS — real transcranial direct current stimulation,10 sessions, 2mA for 20 minutes
  Arms: Verum tDCS; real VRT
Device: sham tDCS — sham transcranial direct current stimulation, 10 sessions, for 20 minutes
  Arms: real VRT; sham tDCS
Behavioral: VRT — Vision restoration training, 10 sessions, 20 minutes
  Arms: Verum tDCS; sham tDCS

SUMMARY:
The purpose of this Study is to determine whether non-invasive transcranial direct current stimulation (tDCS) is effective in increasing rehabilitation effects after stroke in visual Cortex.

DETAILED DESCRIPTION:
Visual field defects after posterior cerebral artery stroke can be improved by vision restoration training (VRT), but when combined with transcranial direct current stimulation (tDCS) which alters brain excitability, vision restoration can be potentiated in the chronic stage. Because it is possible that such therapy may be more effective during the early recovery phase after the stroke and can reach patients during the rehabilitation phase, investigators wished to explore the applicability, efficacy and safety of early intervention with a combined tDCS/VRT treatment.

19 post-acute stroke homonymous hemianopia patients were randomly assigned to either 10 sessions of combined rea-tDCS (2mA, 10 daily sessions of 15-20 min) and VRT, or sham-tDCS and VRT. The primary outcome criterion was the pre-post change in perimetric detection thresholds. Secondary outcome is neurophysiological changes in EEG measures (VEP, Connectivity, Spectral Power, ...)

ELIGIBILITY:
Inclusion Criteria:

* Posterior Cerebral Artery Stroke
* Visual Field Defect
* Lesion age 4 weeks up to 6 month max.

Exclusion Criteria:

* Electrical Implants
* Metal artefacts in head
* Epilepsy
* Visual Neglect

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change of mean sensitivity (in dB) detection threshold from baseline to post-intervention and follow up | 14-20 days post treatment, 3 months follow up

SECONDARY OUTCOMES:
Change in power spectra (Volts-squared per Hz (V^2/Hz) from baseline to post-intervention and follow up | 14-20 days post treatment, 3 months follow up
  power spectra (Volts-squared per Hz (V^2/Hz)
Change in VEP latencies (ms) from baseline to post-intervention and follow up | 14-20 days post treatment, 3 months follow up
  VEP latencies (ms)
Change in VEP amplitudes (µV) from baseline to post-intervention and follow up | 14-20 days post treatment, 3 months follow up
  VEP amplitudes (µV)
Change in network coherence from baseline to post-intervention and follow up | 14-20 days post treatment, 3 months follow up
  network coherence correlations
Number of participants with treatment-related adverse events assessed by a questionnaire | up to 4 months
  questionnaire recording adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard A Sabel, Prof. Dr., Study Director — Institute of Medical Psychology
Locations (2):
- Neurologisches Therapiezentrum Gmundnerberg, Altmünster, Austria
- Inst. f. Medical Psychology, Univ. of Magdeburg, Magdeburg, Germany

IPD SHARING:
Plan to Share IPD: No